CLINICAL TRIAL: NCT06359275
Title: A Phase II Study on the Safety and Efficacy of PD-1 Combined With Nab-paclitaxel/Gemcitabine and PULSAR in the Treatment of Locally Advanced Unresectable Pancreatic Cancer and Local Recurrence After Surgery.
Brief Title: PD-1 Combined With Chemotherapy and PULSAR in LAPC and Local Recurrence Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iPULSAR-PC
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Immunotherapy; 130-nm albumin-bound paclitaxel; Drug Therapy; Gemcitabine; DEAE-Dextran; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 Combined With chemotherapy + PULSAR. (Experimental): Toripalimab: 240 mg/time, intravenously infused over 30 minutes， administered once every three weeks until the treatment termination event specified in the protocol occurs.
  Paclitaxel for injection (albumin-bound): 125 mg/m2 and infuse intravenously for at least 30 minutes: D1, 8 days of administration. Every 21 days is a cycle.
  Gemcitabine hydrochloride for injection: 1000 mg/m2 for intravenous infusion over 30 minutes: D1, 8 days of administration. Every 21 days is a cycle.
  PULSAR: Hypofractionated or stereotactic radiotherapy for the primary pancreatic tumor lesions and surrounding metastatic lymph nodes, 5-10 Gy/time, in conjunction with the chemotherapy cycle, completed once within each chemotherapy cycle, for a total of 5 times.
  Interventions: Drug: PD-1; Drug: Nab-paclitaxel; Drug: Gemcitabine; Radiation: PULSAR

INTERVENTIONS:
Drug: PD-1 — Toripalimab，240 mg/time，D1， Q3W
  Other Names: immunotherapy
Drug: Nab-paclitaxel — Nab-paclitaxel, 125mg/m2，IV，D1，8, Q3W
  Other Names: chemotherapy
Drug: Gemcitabine — Gemcitabine，1000mg/m2，IV，D1，8，Q3W
  Other Names: chemotherapy
Radiation: PULSAR — 5-10 Gy per session, a total of 5 times.
  Other Names: radiotherapy

SUMMARY:
This trial is a phase II clinical trial of the safety and efficacy of PD-1 antibody (Toripalimab) in combination with paclitaxel (albumin-bound type) and gemcitabine and PULSAR radiotherapy in patients with locally advanced unresectable pancreatic cancer and patients with only local recurrence after pancreatic cancer surgery, to observe the safety and efficacy of PD-1 antibody (Toripalimab) in combination with paclitaxel (albumin-bound type) and gemcitabine and PULSAR in the treatment of patients with locally advanced unresectable pancreatic cancer.

DETAILED DESCRIPTION:
This trial is a phase II clinical trial of the safety and efficacy of PD-1 antibody (Toripalimab) in combination with paclitaxel (albumin-bound type) and gemcitabine and PULSAR radiotherapy in patients with locally advanced unresectable pancreatic cancer and patients with only local recurrence after pancreatic cancer surgery, to observe the safety and efficacy of PD-1 antibody (Toripalimab) in combination with paclitaxel (albumin-bound type) and gemcitabine and PULSAR in the treatment of patients with locally advanced unresectable pancreatic cancer.

Progression-free survival (PFS), objective response rate (ORR), overall survival (OS), surgical conversion rate, and quality of life were observed in subjects with locally advanced unresectable pancreatic cancer with precise histological or cytological diagnosis and patients with only local recurrence after surgery. This is a single-center study. A total of 46 subjects with locally advanced unresectable pancreatic cancer and 35 subjects with locally recurrent pancreatic cancer after surgery were planned to be enrolled.

The estimated enrollment time is 18 months, with at least 18 months of follow-up for each subject.

This trial will evaluate the safety data of all subjects who have received at least one dose of study treatment for analysis. The National Cancer Institute (NCI) Common Adverse Event Evaluation Criteria (CTCAE version 5.0) were used. The efficacy evaluation was done according to the clinical diagnosis and treatment routine-follow-up patients combined with follow-up records.

ELIGIBILITY:
Inclusion Criteria

1. Sign the informed consent form. The subject has received a full explanation and understanding of the purpose, content, predicted efficacy, pharmacological effects, and risks of this trial, and the subject has signed an informed consent form;
2. Target group

   1. Locally advanced pancreatic adenocarcinoma confirmed by histopathology or cytology, or pancreatic cancer with only local recurrence but no distant metastasis after surgery (local recurrence includes tumor bed recurrence and regional lymph node metastasis, which needs to be confirmed by biopsy pathology or PET -CT shows high metabolic activity, more than 6 months after the completion of postoperative adjuvant treatment);
   2. There is at least one measurable objective lesion according to RECIST1.1 standards;
   3. ECOG score 0-1 points;
   4. Expected survival time ≥ 3 months;
   5. Willing to comply with research procedures and able to undergo treatment (including surgery) and follow-up;
   6. There are no contraindications for the use of PD-1, PD-L1, gemcitabine and paclitaxel for injection (albumin-bound);
   7. There are no contraindications to radiotherapy;
3. Abnormal physical examination and laboratory test results

   1. Hematological dysfunction is defined as i) absolute neutrophil (ANC) count ≥1.5×109/L; ii) platelet (PLT) count: ≥80×109/L; iii) hemoglobin (Hb) level ≥ 90g/L.
   2. Abnormal liver function is defined as: i) Total bilirubin (TBil) level: ≤ 1.5 times the upper limit of normal (ULN); ii) Aspartate aminotransferase (AST) and alanine; aminotransferase (ALT) levels ≤ 2.5 times the ULN, if liver metastasis is present, ≤5 times ULN;
   3. Abnormal renal function definition: serum creatinine ≤ 1.5 times ULN, or calculated creatinine clearance ≥ 50ml/min;
   4. Definition of abnormal coagulation function: international normalized ratio (INR) ≤ 1.5 times ULN, and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN, unless the subject is receiving anti- Coagulation treatment.
4. Subjects who are positive for hepatitis B surface antigen (HBsAg) and whose peripheral blood hepatitis B virus deoxyribonucleic acid (HBV-DNA) titer is ≤1×103 copy number/L; if they are HBsAg-positive and whose peripheral blood HBV-DNA titer is detected ≥1×103 copy number/L, if the researcher believes that the subject's chronic hepatitis B is in a stable phase and will not increase the subject's risk, the subject is eligible for inclusion;
5. Age and reproductive status

   1. Men and women aged 18-75;
   2. Subjects of childbearing age must agree to take adequate contraceptive measures during the trial; the serum or urine pregnancy test of women of childbearing age must be negative 24 hours before the start of chemotherapy;
   3. Women must be non-lactating.

Exclusion criteria

1. Have received anti-PD-1 or anti-PD-L1 antibody treatment in the past;
2. Have received any investigational drugs within 4 weeks before using the investigational drugs for the first time;
3. Enroll in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up;
4. Have received radiotherapy for the upper abdomen in the past;
5. Medical history and concurrent diseases

   1. Uncontrolled serious medical diseases that the researcher believes will affect the subject's ability to receive the treatment of the research plan, such as combined with serious medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, and uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc;
   2. Have active, known, or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, hypothyroidism, and need for bronchodilators treatment of asthma, etc.). Subjects with hypothyroidism requiring only hormone replacement therapy and skin diseases not requiring systemic treatment (such as vitiligo, psoriasis, or alopecia) were eligible;
   3. Have active tuberculosis infection. Patients with active pulmonary tuberculosis infection within 1 year before the medication will be excluded, even if they have been treated; patients with a history of active pulmonary tuberculosis infection more than one year ago will also be excluded unless it is proven that they have previously received standard anti-tuberculosis treatment;
   4. Previous interstitial lung disease or (non-infectious) pneumonia requiring oral or intravenous steroid therapy;
   5. Long-term systemic corticosteroids (dose equivalent to >10 mg prednisone/day) or any other form of immunosuppressive treatment are required. Subjects using inhaled or topical corticosteroids were eligible;
   6. Heart disease that is not well controlled, such as:

      1. New York Heart Association (NYHA) grade 2 or above heart failure
      2. Unstable angina pectoris
      3. Myocardial infarction occurred within 1 year
      4. Supraventricular or ventricular arrhythmias that are clinically significant and require treatment or intervention;
   7. Dementia, altered mental status, or any mental illness that would prevent understanding or giving informed consent or completing questionnaires;
   8. History of allergy or hypersensitivity reaction to any component of the treatment;
   9. Malignant tumors within 5 years, except for fully treated basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery;
   10. Previous systemic treatment for locally advanced pancreatic cancer;
   11. Subjects who have been pathologically diagnosed with squamous cell carcinoma (not limited to organs) and received taxane-containing regimens as neoadjuvant/adjuvant treatment;
   12. Subjects with ≥ grade 2 peripheral neuropathy according to CTCAE version 5.0.
6. Hepatitis C virus (HCV) antibody positive or human immunodeficiency virus (HIV) antibody positive;
7. Active infection requiring systemic treatment;
8. Need to be combined with other anti-tumor drug treatments;
9. Have received any experimental drug treatment or participated in another interventional clinical trial within 30 days of the screening period;
10. The researcher believes that other circumstances are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to approximately 1 years
  PFS is defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to approximately 1 years
  ORR is defined as the percentage of subjects with complete response (CR) or partial response (PR) by investigator assessment per RECIST criteria, version 1.1.
Overall survival (OS) | up to approximately 1 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Surgical Conversion Rate | 18 weeks
  The surgery is scheduled to take place after a minimum of 4 weeks from the last dose to allow the effects of the drug to wear off. The eligible subjects can undergo surgery within 8 weeks from the last dose. A successful resection is achieved when a patient achieves R0 or R1 resection. However, if a patient has R2 resection or unresectable, then it is considered as resection failure. The pathology committee of our center determines the surgical results of R0, R1, and R2 based on the tissue obtained during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Weijing Zhang, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanhai, China

IPD SHARING:
Plan to Share IPD: No